CLINICAL TRIAL: NCT02116335
Title: Endothelin Receptor Function and Acute Stress (End-Stress)
Brief Title: Endothelin Receptor Function and Acute Stress
Acronym: End-Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Harris, Assistant Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: End-Stress; 5P01HL069999 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
Keywords: arterial stiffness; flow-mediated dilation; endothelial function; pulse wave velocity; inflammation; oxidative stress; Nitric Oxide; Cold Pressor Test; physio flow; Bosentan; Endothelin Receptor; Endothelin-1; BMI; stress; blood pressure
MeSH Terms: conditions — Hypertension; Inflammation | interventions — Bosentan; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan (Experimental): Sub-Chronic (3 days) Bosentan 250mg/day.
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator): Stress response and endothelial function will be determined following a three day treatment of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — Stress response and vascular function will be assessed 3 days following 125 mg twice per day of Bosentan
  Other Names: Tracleer
  Arms: Bosentan
Drug: Placebo — Stress response and vascular function will be assessed 3 days following twice per day placebo
  Other Names: lactose capsule
  Arms: Placebo

SUMMARY:
Our bodies respond differently to stress. Animal studies by the investigators have found that endothelin-1 plays a role in regulating blood pressure in response to stress. This study is an extension of the investigators previous animal work to evaluate the role of endothelin-1 during stress in humans.

DETAILED DESCRIPTION:
Using a salt sensitive animal model of prehypertension, the Dahl S rat,the investigators have previously published that acute stress elicits a pressor response that is accompanied by an increase in 8 isoprostane and endothelin-1. However, the pressor response is suppressed by endothelin A/B receptor antagonism. Moreover, the investigators have identified that the increase in 8-isoprostane occurs downstream of endothelin receptor activation. These data indicate that endothelin receptor activation is a main player In the pressor response to acute stress in pre-hypertensive animals; however, this phenomenon has yet to be elucidated in humans.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopausal women (Ages 18-50 years old)
* Self-reported Black and White adults
* Lean adults (BMl <25 kg/m^)
* Obese adults (BMl > 30 kg/m^)

Exclusion Criteria:

* Having a BMI less than 16 kg/m2 (severely and very severely underweight) or that is greater than 40 kg/m2 (Class III obesity)
* Having evidence of cardiovascular, pulmonary, renal, hepatic, cerebral, or metabolic disease
* Having evidence of pregnancy
* Using medications that affect vascular tone (i.e., nitrates, etc.)
* Postmenopausal women
* Uncontrolled hypertension
* Individuals who are on a restricted salt diet
* Having a history of chronic pain
* Having a history of rheumatoid arthritis
* Using medications that are contraindicated with bosentan (i.e. glyburide, cyclosporine)
* Liver dysfunction (which may be identified with the blood sample we take)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-06; Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Flow-Mediated Dilation (FMD) | Baseline and 3 days
  Brachial artery FMD induced by reactive hyperemia will be used to assess vascular endothelial function.

SECONDARY OUTCOMES:
Arterial Stiffness Evaluation (PWV) | Baseline and 3 days
  A tonometer will be gently applied on the carotid artery and then the femoral artery and the radial artery to record how fast blood flows between each of the points.
Physio Flow | Baseline and 3 days
  Six surface electrodes will be placed on the body. 2 on the neck, 2 on the chest, and 2 on the back in order to measure parameters of the heart during exercise.
Femoral blood flow | Baseline and 3 days
  Though ultrasound assessment; resistance of the blood flow, blood flow, blood velocity, and arterial diameter will all be measured in the femoral artery during the physically induced stress test which involves submerging the subjects hand in ice water for 3 minutes.
Blood Pressure | Baseline and 3 days
  Blood pressure will measured in response to the physically induced stress test which involves submerging the subjects hand in ice water for 3 minutes.
Resting Energy Expenditure | Baseline and 3 days
  REE will be assessed before and following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, Ph.D., Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Laboratory of Integrative Vascular and Exercise Physiology — http://www.livep.net